CLINICAL TRIAL: NCT03878706
Title: The Effect of GLP-1 Agonist, SGLT2 Inhibitor and Their Combination on Endothelial Function, Arterial Stiffness and Left Ventricular Deformation in Patients With Type 2 Diabetes With High Cardiovascular Risk
Brief Title: The Cardiovascular Effect of GLP-1 Agonist, SGLT2 Inhibitor and Their Combination
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Professor of Cardiology, University of Athens
Other Study IDs: 2790/03-11-2017
Record Dates: First submitted 2019-02-11; First posted 2019-03-18 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Endothelial glycocalyx integrity; Oxidative stress biomarkers; Arterial stiffness; GLS; NT-proBNP; GDF-15; MOTS-c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — Blood sample obtained from the subjects for oxidative stress markers (malondialdehyde and protein carbonyls), vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15 and mitochondrial-derived peptide-c (MOTS-c) measuring.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GLP1 and SGLT2i group: 60 patients treated with a combination of liraglutide and empagliflozin. All subjects will undergo an echocardiographic study to estimate GLS, left ventricular twisting-untwisting using speckle tracking imaging and carotid intima-media thickness. PWV, AIx, SBPao and PPao with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of sublingual vessels using Sideview Darkfield Imaging (Microscan, Glycockeck). PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx. Oxidative stress markers, vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15, mitochondrial-derived peptide-c (MOTS-c), blood glucose, glycosylated hemoglobin (HbA1c) and lipid profile will be measured before and at 6 and 12 months of treatment.
- GLP1 group: 60 patients treated with liraglutide. All subjects will undergo an echocardiographic study in order to estimate GLS, left ventricular twisting-untwisting using speckle tracking imaging and carotid intima-media thickness. PWV, AIx, SBPao and PPao with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of sublingual vessels using Sideview Darkfield Imaging (Microscan, Glycockeck). PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx. Oxidative stress markers, vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15, mitochondrial-derived peptide-c (MOTS-c), blood glucose, glycosylated hemoglobin (HbA1c) and a full lipidemic profile will be measured before and at 6 and 12 months of treatment.
- SGLT2i group: 60 patients treated with empagliflozin. All subjects will undergo an echocardiographic study in order to estimate GLS, left ventricular twisting-untwisting using speckle tracking imaging and carotid intima-media thickness. PWV, AIx, SBPao and PPao with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of sublingual vessels using Sideview Darkfield Imaging (Microscan, Glucockeck). PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx. Oxidative stress markers, vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15, mitochondrial-derived peptide-c (MOTS-c), blood glucose, glycosylated hemoglobin (HbA1c) and a full lipidemic profile will be measured before and at 6 and 12 months of treatment.
- Control group: 60 patients treated with insulin and metformin.All subjects will undergo an echocardiographic study in order to estimate GLS, left ventricular twisting-untwisting using speckle tracking imaging and carotid intima-media thickness. PWV, AIx, SBPao and PPao with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of subglottic vessels using Sideview Darkfield Imaging (Microscan, Glucockeck). PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx. Oxidative stress markers, vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15, mitochondrial-derived peptide-c (MOTS-c), blood glucose, glycosylated hemoglobin (HbA1c) and a full lipidemic profile will be measured before and at 6 and 12 months of treatment.

SUMMARY:
A. Four groups of patients with type 2 diabetes mellitus with high or very high cardiovascular risk or heart failure with preserved ejection fraction (HFpEF) will be studied before and at 6 and 12 months of treatment:

* 60 patients treated with a combination of GLP1 analogue and SGLT2 inhibitor ± metformin
* 60 patients treated with GLP-1 agonist as a second step after metformin
* 60 patients treated with SGLT2 inhibitor as a second step after metformin
* 60 patients treated with a combination of insulin and other antidiabetic agents (metformin - DPP4 inhibitors) Individuals will be equal distributed as far as age, gender and body mass index concerned. In addition, patients suffered from kidney disease and retinopathy are excluded.

DETAILED DESCRIPTION:
Disordered glucose tolerance in patients with type 2 diabetes mellitus is multifactorial and includes dysfunction not only of β-cells of the pancreas, liver and muscles, but also of the adipose tissue, gastrointestinal tract, kidney, α-cells of the pancreas and the brain. Therefore, it is likely that the use of drugs that act on multiple aspects of the pathophysiology of diabetes will have beneficial effects on glycemic control and outcome of patients.In addition to the many possible causes of glucose deregulation, people with type 2 diabetes have comorbidities such as hypertension, hyperlipidemia and obesity resulting in increased cardiovascular risk. Optimal treatment of hyperglycaemia and cardiovascular risk factors is necessary to reduce adverse events. Although the initial approach is the modification of dietary factors (physical activity, diet, smoking cessation), the progressive nature of type 2 diabetes ultimately leads to the use of multiple therapies. Guidelines for the treatment of patients with type 2 diabetes with high HbA1c are initial double-combined therapy or triple combination if glycemic control is not achieved after 3 months. Although insulin is usually included in such combinations, additional treatment options are required for patients with high HbA1c who also need to lose weight and avoid hypoglycaemia. It is likely that the outcome of patients could be improved by using drugs targeting different aspects of the disease (glycemia, body weight, blood pressure, lipids).

Over the last decade, two classes of antidiabetic drugs have been added to weight loss, improved cardiovascular risk factors and a low risk of hypoglycemia: glucagon-like peptide-1 agonists (GLP-1, glucagon like peptide-1) and inhibitors of the sodium glucose subtype 2 (SGLT2, sodium-glucose co-transporters). Recent studies have shown that these two drugs have cardioprotective effects possibly through different mechanisms of action, while their complementary mechanical, pharmacological and clinical effects make their combination (in addition to metformin) potentially beneficial in type 2 diabetes patients. Specifically, SGLT2 inhibitors manifest their cardioprotective activity by improving hemodynamic parameters, while GLP-1 agonists through antiatherogen / anti-inflammatory mechanisms.

The increased arterial stiffness with the associated increase in the range of reflected pressure waves, determines not only the augmentation of systolic pressure but also the rate of increase which depends on age. Increased levels of pulse pressure (indirect atherosclerotic index) and pulse wave velocity (PWV), a reliable measure of arterial stiffness, predict future cardiovascular events. Endothelial dysfunction is associated with the presence of atherosclerosis and is also considered as an indicator of the early changes preceding it. The role of impaired endothelial function of large arteries seems to be significant in the pathogenesis of cardiovascular disease. Endothelial glycocalyx is a glycoprotein layer that covers the surface of endothelial cells and regulates arterial wall permeability and the interaction of endothelial cells with circulating blood cells. Inflammatory or atherogenic stimuli, such as hyperglycemia, lead to glucocalyx disorder and increased vascular sensitivity to further atherogenic stimuli. The two-dimensional speckle tracking ultrasound allows accurate estimation of left ventricular distortion, which is disordered in diabetics in relation to healthy subjects.

Hypothesis of the proposed study:

Endothelial function, arterial stiffness and left ventricular deformation are improved in patients with type 2 diabetes with high or very high cardiovascular risk or heart failure with preserved ejection fraction (HFpEF) treated with GLP-1 agonist and SGLT2 inhibitor compared to either one or both combination of insulin and other antidiabetic tablets.

Aim of the study:

The aim of this study is to investigate the effect of GLP-1 agonist, SGLT2 inhibitor and their combination on endothelial function, arterial stiffness, central hemodynamic characteristics and left ventricular deformation in patients with type 2 diabetes with high or very high cardiovascular risk or HFpEF and compared with the combination of insulin and other antidiabetic tablets.

Materials and methods :

A. Four groups of patients with type 2 diabetes mellitus with high or very high cardiovascular risk or HFpEF will be studied before and at 6 and 12 months of treatment:

* 60 patients treated with a combination of GLP1 analogue and SGLT2 inhibitor ± metformin
* 60 patients treated with GLP-1 agonist as a second step after metformin
* 60 patients treated with SGLT2 inhibitor as a second step after metformin
* 60 patients treated with a combination of insulin and other antidiabetic agents (metformin - DPP4 inhibitors) Individuals will be equal distributed as far as age, gender and body mass index concerned. In addition, patients suffered from kidney disease and retinopathy are excluded.

B. All patients will be submitted to an echocardiographic study in order to estimate the total left ventricular and atrial myocardial global longitudinal strain (GLS) as well as the twisting-untwisting of the left ventricle using speckle tracking imaging. In addition, pulse wave velocity (PWV, measured in m/s), pulse wave augmentation index [AIx %, which is calculated by the formula (P2-P1)/PP x 100, where P1 stands for peak systolic pressure, P2 stands for second peak systolic pressure due to wave reflection and PP stands for Pulse Pressure], central systolic blood pressure (SBPao, measured in mm Hg) and central pulse pressure (PPao, measured in mm Hg) with Arteriograph, Mobilograph and Complior, and perfused boundary region (PBR) of sublingual vessels (5-25 μm in size) using a high-resolution camera with Sideview Darkfield Imaging technique (Microscan, Glucockeck). PBR consists the cell-free space which is formed from the separation of red blood cells from plasma at the surface of the endothelial glycocalyx. Increased PBR is considered to be an accurate indicator of the reduction of endothelial glycocalyx thickness due to plasma penetration into the glycocalyx.

Μalondialdehyde (MDA), protein carbonyls (PC) as oxidative stress markers, vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates, N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15, mitochondrial-derived peptide-c (MOTS-c), blood glucose, glycosylated hemoglobin HbA1c and a full lipidemic profile will be measured before and at 6 months and at 12 months of treatment.

The examination will be carried out at the Laboratory of Preventive Cardiology of the 2nd Department of Cardiology of the University of Athens at "Attikon" Hospital. Τhe investigators will also compare the participants with history of coronary artery disease with those without hisotry of coronary artery disease.

C. For the statistical analysis of the results, the significance of each intervention will be measured by t-test and the 4 groups will be compared by ANOVA (post-hoc comparisons with Bonferroni correction). Non-parametric tests will be used for non-Gaussian distributions. Forty individuals should be included in each group in order the results being statistically significant. In a previous study, myocardial global longitudinal strain of the left ventricle showed normal distribution with standard deviation 10. A true difference in mean left ventricular myocardial distortion between the intervention group (GLP-1 agonist compined with SGLT2 inhibitor) and a control one (combination of insulin and other antidiabetic tablets) which is calculated of -6.344% or 6.344% will be calculated with probability 0.8. The probability of a type I error if the null hypothesis is that the mean difference between the two groups is equal, is equivalent to 0.05.

Significance/future prospects:

This study is expected to open the horizons of better understanding the cardiovascular benefits of GLP-1 agonist, SGLT2 inhibitor and their combination in patients with type 2 diabetes mellitus. Moreover, the contribution of the investigator's results, in a clinical-level could be the use of new drug therapies that reduce both microvascular complications by reducing glycemia and macrovascular complications (myocardial infarction, stroke, cardiovascular mortality) as the first treatment line in patients with type 2 diabetes with high or very high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Subject has type 2 diabetes mellitus
* Subject has high or very high cardiovascular risk
* Subject has heart failure with preserved ejection fraction

Exclusion Criteria:

* Subject has type 1 diabetes mellitus
* Subject has kidney disease
* Subject has retinopathy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 240 individuals (60 subjects in each group)
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of Global Longitudinal Strain (GLS) difference among treatment groups. | 12 months
  Comparison of Global Longitudinal Strain (GLS) difference among treatment groups, measured by echocardiographic study

SECONDARY OUTCOMES:
Comparison of arterial stiffness markers difference among treatment groups. | 12 months
  Comparison of pulse wave velocity difference among treatment groups
Comparison of wave reflection markers difference among treatment groups | 12 months
  Comparison of central augmentation index (Aix%) difference among treatment groups
Comparison of central aortic blood pressure differences among treatment groups | 12 months
  Comparison of both central systolic and diastolic aortic blood pressure differences among treatment groups
Comparison of endothelial glycocalyx thickness difference among treatment groups | 12 months
  Comparison of Perfused Boundary Region (PBR) difference of sublingual vessels among treatment groups
Comparison of oxidative stress and endothelial function biomarkers differences among treatment groups | 12 months
  Comparison of malondialdehyde, protein carbonyls vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates plasma levels differences among treatment groups
Comparison of cardiac biomarkers differences among treatment groups. | 12 months
  Comparison of N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15 and mitochondrial-derived peptide-c (MOTS-c) levels differences among treatment groups
Comparison of left ventricular myocardial function difference between coronary artery disease patients and non-coronary artery disease patients in each study group. | 12 months
  Comparison of Global Longitudinal Strain (GLS) difference between coronary artery disease patients and non-coronary artery disease patients in each study group.
Comparison of arterial stiffness difference between coronary artery disease patients and non-coronary artery disease patients in each study group. | 12 months
  Comparison of pulse wave velocity difference between coronary artery disease patients and non-coronary artery disease patients in each study group.
Comparison of endothelial glycocalyx thickness difference between coronary artery disease patients and non-coronary artery disease patients in each study group. | 12 months
  Comparison of Perfused Boundary Region (PBR) difference between coronary artery disease patients and non-coronary artery disease patients in each study group.
Comparison of oxidative stress and endothelial function biomarkers differences between coronary artery disease patients and non-coronary artery disease patients in each study group. | 12 months
  Comparison of malondialdehyde, protein carbonyls, vascular cell adhesion molecule (VCAM)-1, intercellular adhesion molecule (ICAM)-1, thrombomodulin, nitrites and nitrates plasma levels difference between coronary artery disease patients and non-coronary artery disease patients in each study group.
Comparison of cardiac biomarkers differences between coronary artery disease patients and non-coronary artery disease patients in each study group. | 12 months
  Comparison of N-terminal pro B-type natriuretic peptide (NT-proBNP), growth differentiation factor (GDF)-15 and mitochondrial-derived peptide-c (MOTS-c) levels difference between coronary artery disease patients and non-coronary artery disease patients in each study group.
Comparison of liver steatosis level between treatment groups | 12 months
  Comparison of Fibrosis-4 (FIB-4) Index for Liver Fibrosis and Non Alcoholic Fatty Liver Disease Score between treatment groups
Comparison of carotid atherosclerotic markers between treatment groups | 12 months
  Comparison of carotid intima-media thickness between treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, Prof, Principal Investigator — 2nd Department of Cardiology, National and Kapodistrian University of Athens; Aimilianos N. Kalogeris, MD, Principal Investigator — 2nd Department of Cardiology, University of Athens; John A. Thymis, MD, Principal Investigator — 2nd Department of Cardiology,University of Athens; Vaia Lambadiari, Prof., Principal Investigator — National and Kapodistrian University of Athens; Georgios Dimitriadis, Prof., Study Chair — National and Kapodistrian University of Athens; Efstathios Iliodromitis, Prof., Study Chair — National and Kapodistrian University of Athens
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Handelsman Y, Bloomgarden ZT, Grunberger G, Umpierrez G, Zimmerman RS, Bailey TS, Blonde L, Bray GA, Cohen AJ, Dagogo-Jack S, Davidson JA, Einhorn D, Ganda OP, Garber AJ, Garvey WT, Henry RR, Hirsch IB, Horton ES, Hurley DL, Jellinger PS, Jovanovic L, Lebovitz HE, LeRoith D, Levy P, McGill JB, Mechanick JI, Mestman JH, Moghissi ES, Orzeck EA, Pessah-Pollack R, Rosenblit PD, Vinik AI, Wyne K, Zangeneh F. American association of clinical endocrinologists and american college of endocrinology - clinical practice guidelines for developing a diabetes mellitus comprehensive care plan - 2015. Endocr Pract. 2015 Apr;21 Suppl 1(Suppl 1):1-87. doi: 10.4158/EP15672.GL. No abstract available. PMID 25869408
- [Result] American Diabetes Association. 7. Approaches to Glycemic Treatment. Diabetes Care. 2016 Jan;39 Suppl 1:S52-9. doi: 10.2337/dc16-S010. No abstract available. PMID 26696682
- [Result] Jabbour SA, Hardy E, Sugg J, Parikh S; Study 10 Group. Dapagliflozin is effective as add-on therapy to sitagliptin with or without metformin: a 24-week, multicenter, randomized, double-blind, placebo-controlled study. Diabetes Care. 2014;37(3):740-50. doi: 10.2337/dc13-0467. Epub 2013 Oct 21. PMID 24144654
- [Result] Nauck MA, Kemmeries G, Holst JJ, Meier JJ. Rapid tachyphylaxis of the glucagon-like peptide 1-induced deceleration of gastric emptying in humans. Diabetes. 2011 May;60(5):1561-5. doi: 10.2337/db10-0474. Epub 2011 Mar 23. PMID 21430088
- [Result] Shaefer CF Jr, Kushner P, Aguilar R. User's guide to mechanism of action and clinical use of GLP-1 receptor agonists. Postgrad Med. 2015;127(8):818-26. doi: 10.1080/00325481.2015.1090295. Epub 2015 Sep 15. PMID 26371721
- [Result] van Bloemendaal L, Ten Kulve JS, la Fleur SE, Ijzerman RG, Diamant M. Effects of glucagon-like peptide 1 on appetite and body weight: focus on the CNS. J Endocrinol. 2014 Mar 7;221(1):T1-16. doi: 10.1530/JOE-13-0414. Print 2014 Apr. PMID 24323912
- [Result] Wanner C, Inzucchi SE, Lachin JM, Fitchett D, von Eynatten M, Mattheus M, Johansen OE, Woerle HJ, Broedl UC, Zinman B; EMPA-REG OUTCOME Investigators. Empagliflozin and Progression of Kidney Disease in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):323-34. doi: 10.1056/NEJMoa1515920. Epub 2016 Jun 14. PMID 27299675
- [Result] Ferrannini G, Hach T, Crowe S, Sanghvi A, Hall KD, Ferrannini E. Energy Balance After Sodium-Glucose Cotransporter 2 Inhibition. Diabetes Care. 2015 Sep;38(9):1730-5. doi: 10.2337/dc15-0355. Epub 2015 Jul 15. PMID 26180105
- [Result] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Result] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Result] Frias JP, Guja C, Hardy E, Ahmed A, Dong F, Ohman P, Jabbour SA. Exenatide once weekly plus dapagliflozin once daily versus exenatide or dapagliflozin alone in patients with type 2 diabetes inadequately controlled with metformin monotherapy (DURATION-8): a 28 week, multicentre, double-blind, phase 3, randomised controlled trial. Lancet Diabetes Endocrinol. 2016 Dec;4(12):1004-1016. doi: 10.1016/S2213-8587(16)30267-4. Epub 2016 Sep 16. PMID 27651331
- [Result] Chae CU, Pfeffer MA, Glynn RJ, Mitchell GF, Taylor JO, Hennekens CH. Increased pulse pressure and risk of heart failure in the elderly. JAMA. 1999 Feb 17;281(7):634-9. doi: 10.1001/jama.281.7.634. PMID 10029125
- [Result] Franklin SS, Khan SA, Wong ND, Larson MG, Levy D. Is pulse pressure useful in predicting risk for coronary heart Disease? The Framingham heart study. Circulation. 1999 Jul 27;100(4):354-60. doi: 10.1161/01.cir.100.4.354. PMID 10421594
- [Result] Domanski M, Norman J, Wolz M, Mitchell G, Pfeffer M. Cardiovascular risk assessment using pulse pressure in the first national health and nutrition examination survey (NHANES I). Hypertension. 2001 Oct;38(4):793-7. doi: 10.1161/hy1001.092966. PMID 11641288
- [Result] Laurent S, Boutouyrie P, Asmar R, Gautier I, Laloux B, Guize L, Ducimetiere P, Benetos A. Aortic stiffness is an independent predictor of all-cause and cardiovascular mortality in hypertensive patients. Hypertension. 2001 May;37(5):1236-41. doi: 10.1161/01.hyp.37.5.1236. PMID 11358934
- [Result] Meaume S, Benetos A, Henry OF, Rudnichi A, Safar ME. Aortic pulse wave velocity predicts cardiovascular mortality in subjects >70 years of age. Arterioscler Thromb Vasc Biol. 2001 Dec;21(12):2046-50. doi: 10.1161/hq1201.100226. PMID 11742883
- [Result] Avolio AP, Deng FQ, Li WQ, Luo YF, Huang ZD, Xing LF, O'Rourke MF. Effects of aging on arterial distensibility in populations with high and low prevalence of hypertension: comparison between urban and rural communities in China. Circulation. 1985 Feb;71(2):202-10. doi: 10.1161/01.cir.71.2.202. PMID 3965165
- [Result] Vaitkevicius PV, Fleg JL, Engel JH, O'Connor FC, Wright JG, Lakatta LE, Yin FC, Lakatta EG. Effects of age and aerobic capacity on arterial stiffness in healthy adults. Circulation. 1993 Oct;88(4 Pt 1):1456-62. doi: 10.1161/01.cir.88.4.1456. PMID 8403292
- [Result] Ikonomidis I, Lekakis J, Papadopoulos C, Triantafyllidi H, Paraskevaidis I, Georgoula G, Tzortzis S, Revela I, Kremastinos DT. Incremental value of pulse wave velocity in the determination of coronary microcirculatory dysfunction in never-treated patients with essential hypertension. Am J Hypertens. 2008 Jul;21(7):806-13. doi: 10.1038/ajh.2008.172. Epub 2008 May 22. PMID 18497732
- [Result] Tzortzis S, Ikonomidis I, Lekakis J, Papadopoulos C, Triantafyllidi H, Parissis J, Trivilou P, Paraskevaidis I, Anastasiou-Nana M, Kremastinos DT. Incremental predictive value of carotid intima-media thickness to arterial stiffness for impaired coronary flow reserve in untreated hypertensives. Hypertens Res. 2010 Apr;33(4):367-73. doi: 10.1038/hr.2010.2. Epub 2010 Feb 5. PMID 20139923
- [Result] Ikonomidis I, Makavos G, Papadavid E, Varoudi M, Andreadou I, Gravanis K, Theodoropoulos K, Pavlidis G, Triantafyllidi H, Parissis J, Paraskevaidis I, Rigopoulos D, Lekakis J. Similarities in coronary function and myocardial deformation between psoriasis and coronary artery disease: the role of oxidative stress and inflammation. Can J Cardiol. 2015 Mar;31(3):287-95. doi: 10.1016/j.cjca.2014.11.002. Epub 2014 Nov 6. PMID 25660150
- [Result] Ikonomidis I, Pavlidis G, Lambadiari V, Kousathana F, Varoudi M, Spanoudi F, Maratou E, Parissis J, Triantafyllidi H, Dimitriadis G, Lekakis J. Early detection of left ventricular dysfunction in first-degree relatives of diabetic patients by myocardial deformation imaging: The role of endothelial glycocalyx damage. Int J Cardiol. 2017 Apr 15;233:105-112. doi: 10.1016/j.ijcard.2017.01.056. Epub 2017 Jan 8. PMID 28096045
- [Result] Ikonomidis I, Tzortzis S, Tsantes A, Ntai K, Triantafyllidi H, Trivilou P, Katsimaglis G, Dima K, Parissis J, Lekakis J. The interplay between renin-angiotensin system activation, abnormal myocardial deformation and neurohumoral activation in hypertensive heart disease: a speckle tracking echocardiography study. Int J Cardiovasc Imaging. 2017 Mar;33(3):323-329. doi: 10.1007/s10554-016-1010-1. Epub 2016 Oct 27. PMID 27787699
- [Result] Pieske B, Tschope C, de Boer RA, Fraser AG, Anker SD, Donal E, Edelmann F, Fu M, Guazzi M, Lam CSP, Lancellotti P, Melenovsky V, Morris DA, Nagel E, Pieske-Kraigher E, Ponikowski P, Solomon SD, Vasan RS, Rutten FH, Voors AA, Ruschitzka F, Paulus WJ, Seferovic P, Filippatos G. How to diagnose heart failure with preserved ejection fraction: the HFA-PEFF diagnostic algorithm: a consensus recommendation from the Heart Failure Association (HFA) of the European Society of Cardiology (ESC). Eur J Heart Fail. 2020 Mar;22(3):391-412. doi: 10.1002/ejhf.1741. Epub 2020 Mar 5. PMID 32133741
- [Derived] Ikonomidis I, Pavlidis G, Pliouta L, Katogiannis K, Maratou E, Thymis J, Michalopoulou E, Prentza V, Katsanaki E, Vlachomitros D, Kountouri A, Korakas E, Andreadou I, Kouretas D, Parissis J, Lambadiari V. Effects of Glucagon-Like Peptide-1 Receptor Agonists, Sodium-Glucose Cotransporter-2 Inhibitors, and Their Combination on Neurohumoral and Mitochondrial Activation in Patients With Diabetes. J Am Heart Assoc. 2025 Mar 4;14(5):e039129. doi: 10.1161/JAHA.124.039129. Epub 2025 Feb 26. PMID 40008510
- [Derived] Ikonomidis I, Pavlidis G, Thymis J, Birba D, Kalogeris A, Kousathana F, Kountouri A, Balampanis K, Parissis J, Andreadou I, Katogiannis K, Dimitriadis G, Bamias A, Iliodromitis E, Lambadiari V. Effects of Glucagon-Like Peptide-1 Receptor Agonists, Sodium-Glucose Cotransporter-2 Inhibitors, and Their Combination on Endothelial Glycocalyx, Arterial Function, and Myocardial Work Index in Patients With Type 2 Diabetes Mellitus After 12-Month Treatment. J Am Heart Assoc. 2020 May 5;9(9):e015716. doi: 10.1161/JAHA.119.015716. Epub 2020 Apr 24. PMID 32326806